CLINICAL TRIAL: NCT06957626
Title: Development and Validation of Microbiota and Metabolite-based Prediction Model for Recurrence of High-risk Colorectal Polyps After Polypectomy
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Jing-Nan Li, Chief physician, Professor, Peking Union Medical College Hospital
Other Study IDs: I-23PJ699
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Polyp; Colorectal Cancer Recurrent; Colorectal Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who undergo colonoscopy with precence of high-risk colorectal polyps: For patients who undergo colonoscopy with presence of high-risk colorectal polyps, collect 1-2 pieces of large intestinal mucosa of the polyp and the normal appearing mucosa surrounding the polyp. Collect stool samples and baseline information such as age, gender and eating habit.
  Each patient will be followed for 3 years, and colonoscopy will be reviewed to determine the recurrence. Biopsies of large intestinal mucosa and stools will be collected at surveillance colonoscopy (follow-up) if allowed. All the samples are stored at -80°C by the study team until the time of DNA extraction for microbiota sequencing analysis and/or metabolomic analysis.

SUMMARY:
The characteristics of the intestinal microbiota in high-risk colorectal polyp recurrence and their relationship with disease pathogenesis have not yet been fully elucidated. This study aims to analyze the microbial community characteristics in the intestinal mucosal tissue of patients after polypectomy with recurrence of colorectal polyps. Additionally, this research holds significant importance for understanding the etiology of adenoma recurrence and develop a microbiota and metabolite-based predicting tool.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 40-75 years who undergo the colonoscopy with at least 1 advanced premalignant polyps or ≥ 3 adenoma

Exclusion Criteria:

* patient with severe physical diseases that prevented them from adhering to the examination requirements,
* patient with coagulopathy or other contraindications for biopsy or polypectomy,
* patient with previous surgical procedures on the gastrointestinal tract,
* presence of colorectal cancer or other malignant tumor at baseline
* presence of inflammatory bowel disease or hereditary polyposis syndromes (such as family adenomatous polyposis or Lynch syndrome)
* within 1 month before enrollment, oral antibiotics and probiotics were taken;
* inability to provide informed consent or refusal to participate in the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with high-risk colorectal polyps
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
The characteristics of the intestinal microbiota in patients with high-risk colorectal polyp recurrence | 24 months
  Analyze the characteristics of the microbiota within the intestinal mucosal tissue of patients with high-risk colorectal polyp recurrence or without recurrence.

SECONDARY OUTCOMES:
Development and validation of Microbiota and metabolite-based model predicting recurrence of high-risk colorectal polyps after polypectomy | 36 months
  Select the recurrence and non-recurrence of polyps during the follow-up period , and develop and validate the recurrence prediction model according to the differences in intestinal mucosal flora and host gene expression levels.

CONTACTS AND LOCATIONS:
Overall Officials: Jing nan Li, MD, Ph.D, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, 1 Shuaifuyuan, Dongcheng District, Beijing, China, Beijing, China

IPD SHARING:
Plan to Share IPD: No